CLINICAL TRIAL: NCT04714918
Title: Chinese Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD) Prevalence Survey
Brief Title: Chinese CKD-MBD Prevalence Survey (CRISS-MBD)
Status: Recruiting | Type: Observational
Sponsor: Limeng Chen (Other)
Responsible Party: Sponsor-Investigator, Limeng Chen, Deputy Director, Department of Nephrology, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: CRISS-MBD
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Chronic Kidney Diseases; Chronic Kidney Disease-Mineral and Bone Disorder
Keywords: Chronic Kidney Diseases; Chronic Kidney Disease-Mineral and Bone Disorder; Hypocalcemia; Hyperphosphatemia; Secondary Hyperparathyroidism
MeSH Terms: conditions — Renal Insufficiency, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder; Hypocalcemia; Hyperphosphatemia; Hyperparathyroidism, Secondary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-center cross sectional epidemiological study. The purpose of this study is to investigate the prevalence of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD) in Chinese population.

DETAILED DESCRIPTION:
The prevalence of Chronic Kidney Disease (CKD) in Chinese population is over 10% and increasing rapidly. Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD) is a constellation of conditions secondary to CKD, including 1) metabolic disorders of calcium, phosphorus and Parathyroid Hormone (PTH), 2) bone diseases and 3) calcifications in blood vessels and soft tissues. CKD-MBD could increase the risks of cardiovascular diseases and bone fracture and overall mortality. However, the data of prevalence of CKD-MBD in Chinese population with different CKD stages is lacking. This is a multi-center cross sectional epidemiological study. The purpose of this study is to investigate the prevalence of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD) in Chinese population.This is a multi-center cross sectional epidemiological study. The purpose of this study is to investigate the prevalence of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD) in Chinese population. A questionnaire was designed to collect the information of demographic data, medical history, laboratory test results and medications from the patients. Multistage stratified cluster sampling method will be used. Based on the sample size estimation, a total of 14-28 tertiary hospitals and 42-56 level II hospitals distributed in seven different geographic regions across China will be included. At least 9863 subjects will be enrolled. The primary outcome is the prevalence of CKD-MBD, including the prevalence of hypocalcemia, hyperphosphatemia and secondary hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Kidney damage for ≥ 3 months, and one of the following criteria:

  1. Glomerular filtration rate (GFR) <60 mL/min/1.73m2 for 3 months or more, irrespective of cause.
  2. proteinuria (>30 mg of urinary albumin excretion per gram of urinary creatinine, > 50 mg of urinary protein excretion per gram of urinary creatinine, >1+ for proteinuria in dipstick, > 0.3g of 24 hour urine protein)
  3. structural renal abnormalities
* hospitalized patients not on dialysis or dialysis patients followed regularly in Hemodialysis centers or Peritoneal Dialysis centers

Exclusion Criteria:

* no available test results within 3 months prior to this study
* no available information of medication or past medical history

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study plans to include hospitalized CKD patients who are not on dialysis and dialysis patients followed regularly in HD centers or PD centers.
Sampling Method: Probability Sample
Enrollment: 10254 (Estimated)
Dates: Start 2020-11-29 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence of hyperphosphatemia | At the end of the enrollment.
  The prevalence of hyperphosphatemia (serum phosphate > 1.45mmol/L) in the whole study population and in participants with different CKD stages.

SECONDARY OUTCOMES:
The prevalence of hypocalcemia | At the end of the enrollment.
  The prevalence of hypocalcemia (serum calcium < 2.13mmol/L) in the whole study population and in participants with different CKD stages.
The prevalence of secondary hyperparathyroidism | At the end of the enrollment.
  The prevalence of secondary hyperparathyroidism (iPTH > 300pg/ml) in the whole study population and in participants with different CKD stages.
The prevalence of hypercalcemia | At the end of the enrollment.
  The prevalence of hypercalcemia (serum calcium > 2.70mmol/L) in the whole study population and in participants with different CKD stages.
The prevalence of bone fracture | At the end of the enrollment.
  The prevalence of bone fracture in the whole study population and in participants with different CKD stages.
The prevalence of vascular calcification | At the end of the enrollment.
  The prevalence of vascular calcification identified by CT scan or ultrasound in the whole study population and in participants with different CKD stages.

CONTACTS AND LOCATIONS:
Overall Officials: Limeng Chen, MD, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (40):
- China (40):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Lu-He Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Hospital of Fangshan District, Beijing, Beijing, Beijing Municipality
  - Beijing Daxing District People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing Hospital of Traditional Chinese Medicine, Chongqing, Chongqing Municipality
  - The Ninth People's Hospital of Chongqing, Chongqing, Chongqing Municipality
  - The Third Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - People's Hospital of Liangping District, Chongqing, Chongqing, Chongqing Municipality
  - The People's Hospital of Fengdu County, Chongqing, Chongqing Municipality
  - The People's Hospital of Nanchuan District, Chongqing, Chongqing, Chongqing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian
  - Zhangzhou People's Hospital, Zhangzhou, Fujian
  - Shunde Hospital of Southern Medical University, The first People's Hospital of Shunde, Foshan, Guangdong
  - Panyu Central Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The Seventh Affiliated Hospital, Sun Yat-sen University, Shenzhen, Guangdong
  - The People's Hospital of Longhua, The Affiliated Hospital of Southern Medical University, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Third People's Hospital of Yiyang, Yiyang, Hunan
  - Anshan Central Hospital, Lishan District, Anshan, Liaoning
  - Benxi Steel General Hospital of Liaoning Health Industry Group, Benxi, Liaoning
  - Dalian University Affiliated Xinhua Hospital, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Traditional Chinese Hospital of Guyuan, Guyuan, Ningxia
  - People's Hospital of Longde County, Guyuan, Ningxia
  - The Fifth People's Hospital of Ningxia Hui Autonomous Region, Shizuishan, Ningxia
  - People's Hospital of Wuzhong, Wuzhong, Ningxia
  - People's Hospital of Tongxin County, Wuzhong, Ningxia
  - People's Hospital of Yanchi County, Wuzhong, Ningxia
  - People's Hospital of Yuanzhou District, Wuzhong, Ningxia
  - Ningxia Chinese Medicine Research Center, Yinchuan, Ningxia
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - The First People's Hospital of Yinchuan, Yinchuan, Ningxia
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
To comply with laws in China, local regulations and hospital policy, IPD sharing might be restricted.

REFERENCES:
- [Result] Zhou C, Wang F, Wang JW, Zhang LX, Zhao MH. Mineral and Bone Disorder and Its Association with Cardiovascular Parameters in Chinese Patients with Chronic Kidney Disease. Chin Med J (Engl). 2016 Oct 5;129(19):2275-80. doi: 10.4103/0366-6999.190678. PMID 27647184
- [Result] Kong X, Zhang L, Zhang L, Chen N, Gu Y, Yu X, Liu W, Chen J, Peng L, Yuan W, Wu H, Chen W, Fan M, He L, Ding F, Chen X, Xiong Z, Zhang J, Jia Q, Shi W, Xing C, Tang X, Hou F, Shu G, Mei C, Wang L, Xu D, Ni Z, Zuo L, Wang M, Wang H. Mineral and bone disorder in Chinese dialysis patients: a multicenter study. BMC Nephrol. 2012 Sep 21;13:116. doi: 10.1186/1471-2369-13-116. PMID 22994525